CLINICAL TRIAL: NCT05391555
Title: Pupillary Unrest as an Indicator of Central Opioid Effect in Subjects 40-60 Years of Age
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-34917
Record Dates: First submitted 2022-05-13; First posted 2022-05-26 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Opioid Toxicity; Pupillary Miosis; Respiratory Depression
MeSH Terms: conditions — Miosis; Respiratory Insufficiency | interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Remifentanil Infusion and Recovery (Experimental): Participants underwent a 10-minute remifentanil infusion. Pupillary measures were taken a baseline and every 2.5 minutes during the 10-minute infusion and 25-minute recovery period.
  Interventions: Drug: Remifentanil Hydrochloride; Device: Pupillometry measurement

INTERVENTIONS:
Drug: Remifentanil Hydrochloride — Infusion of 0.2 µg/k/m for 5 minutes, the 0.3 µg/k/m for 5 minutes.
Device: Pupillometry measurement — Pupillary measurements were taken at baseline and every 2.5 minutes during the 10-minute infusion and 25-minute recovery period.

SUMMARY:
This study will establish the relationship between magnitude of opioid exposure and a pupillary measure referred to as PUAL (pupillary unrest in ambient light), in subjects aged 40-60. Previous investigation demonstrated that loss of PUAL was a sensitive, discriminative indicator of opioid toxicity and respiratory depression among subjects aged 20-40 years old. Population data indicate that pupil size and PUAL decline slightly with age. The investigators will explore whether PUAL proves to be a sensitive indicator of opioid exposure and respiratory depression in this older group.

DETAILED DESCRIPTION:
Healthy volunteer subjects aged 40-60 will receive a standardized weight-based 10-minute remifentanil infusion protocol to achieve a peak estimated remifentanil effect site concentration of approximately 6 ng/mL. Pupillary measures will be taken at baseline and regular time intervals during and after the infusion, over a period of 35 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, BMI < 35 kg/m2

Exclusion Criteria:

* current or recent opioid use
* opioid or other substance use disorder
* known or suspected OSA or sleep disordered breathing
* ischemic heart disease, heart failure or symptomatic arrhythmia history
* ocular disease or previous eye surgery
* active use of alpha adrenergic blockers, anticholinergic medications,
* active use of antidepressant or mood stabilizing medications
* active use of phosphodiesterase inhibitors
* use of stimulant or appetite suppressant medications
* active use of antihypertensive or antiarrhythmic medications
* use of topical eye medications.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Eshima McKay, MD, Principal Investigator — Professor of Anesthesia
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McKay RE, Kohn MA, Larson MD. Pupillary unrest, opioid intensity, and the impact of environmental stimulation on respiratory depression. J Clin Monit Comput. 2022 Apr;36(2):473-482. doi: 10.1007/s10877-021-00675-3. Epub 2021 Mar 2. PMID 33651243
- [Background] McKay RE, Larson MD. Detection of opioid effect with pupillometry. Auton Neurosci. 2021 Nov;235:102869. doi: 10.1016/j.autneu.2021.102869. Epub 2021 Aug 18. PMID 34474355
- [Background] McKay RE, Neice AE, Larson MD. Pupillary Unrest in Ambient Light and Prediction of Opioid Responsiveness: Case Report on Its Utility in the Management of 2 Patients With Challenging Acute Pain Conditions. A A Pract. 2018 May 15;10(10):279-282. doi: 10.1213/XAA.0000000000000710. PMID 29608463

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remifentanil Infusion and Recovery
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Remifentanil Infusion and Recovery
Number analyzed (Participants) | 10
Age, Customized [Count of Participants; unit: Participants]
  Age 40-60 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White European | 4
  Asian/Pacific Islander | 3
  Black | 1
  Latinx | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Time Concentration Curve (AUROC )
Description: PUAL measured by pupillometer. PUAL at zero-moderate opioid concentration (<1.8 ng/mL) versus high-toxic opioid concentration (>2.5 ng/mL) were dichotomous classifiers.
  Receiver Operating Characteristic curve constructed, with AUROC reported
Time Frame: Baseline, and every 2.5 minutes during 10-minute infusion and 25-minute recovery
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Remifentanil Infusion and Recovery
Number analyzed (Participants) | 10
Probability | 0.9700 [0.9340 to 1.0000]

ADVERSE EVENTS:
Time Frame: 65 minutes.
Arm/Group | Remifentanil Infusion and Recovery
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT05391555/Prot_SAP_000.pdf